CLINICAL TRIAL: NCT05886491
Title: A Phase 1/2a, Open-Label, Dose Escalation, and Dose Expansion Study to Assess the Safety and Efficacy of GDX012 in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Study of GDX012 in Adults With Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-012-1501; jRCT2033240022 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Leukemia
Keywords: Drug Therapy; AML; acute myeloid leukemia; cell therapy; allogenic; gamma delta T cells; relapsed/ refractory
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Dose Escalation of GDX012 (Experimental): Participants will receive GDX012 weight-based dose as intravenous (IV) infusion on Day 1 of Phase 1 after lymphodepleting chemotherapy. Three dose levels of GDX012 will be tested in Phase 1. Some participants may be eligible for a second dose.
  Interventions: Drug: GDX012; Drug: Chemotherapy Agents
- Phase 2a: GDX012 (Experimental): Participants will receive GDX012 (weight-based) IV infusion at pre-selected one or two dose levels from Phase 1, on Day 1 after lymphodepleting chemotherapy. Some participants may be eligible for a second dose.
  Interventions: Drug: GDX012; Drug: Chemotherapy Agents

INTERVENTIONS:
Drug: GDX012 — GDX012 suspension for IV infusion.
Drug: Chemotherapy Agents — Chemotherapy agents (fludarabine/cyclophosphamide) as per standard of care.

SUMMARY:
GDX012 is a novel cell therapy developed for the treatment of certain types of cancer, including Acute Myeloid Leukemia (AML). The main aims of the study are to learn how safe GDX012 is, how treatment with GDX012 is tolerated and to determine the best dose of GDX012.

DETAILED DESCRIPTION:
The drug being tested in this study is called GDX012. GDX012 is being tested to evaluate the safety and tolerability in adult participants with AML.

The study will enroll approximately 53 patients in two phases, dose escalation and dose expansion.

During Phase 1 (sequential dose escalation), participants will be assigned to one of the following treatment groups each consisting of 3 to 6 participants to receive GDX012 at one of the three dose levels:

1. GDX012 Dose 1
2. GDX012 Dose 2
3. GDX012 Dose 3

Upon completion of Phase 1, 1 to 2 dose levels will be selected for Phase 2a of the study. At the completion of Phase 2a of the study a single dose may be selected by the sponsor and investigators as the recommended phase 2 dose (RP2D) for future study.

This multi-center trial will be conducted in the United States. The overall time to participate in the study is approximately 14 months.

ELIGIBILITY:
Inclusion criteria:

1. Total body weight of ≥40 kg.
2. Must have pathologically confirmed relapsed or refractory acute myeloid leukemia (R/R AML) including:

   1. Relapsed AML is defined as ≥5% blasts in the bone marrow (BM) or peripheral blood at any time after achieving a CR, CRh, Cri, or MLFS.
   2. Refractory AML is defined as failure to achieve a CR, CRh, Cri, or MLFS after 1 of the following regimens:

   i. Two courses of intensive induction chemotherapy. ii. At least 2 cycles of hypomethylating agent (HMA) or low-dose, cytarabine-based combination regimen.

   iii. At least 4 cycles of HMA monotherapy.
3. During dose escalation, participants must be ineligible for hematopoietic stem cell transplantation (HSCT).
4. Must have an anticipated life expectancy of >3 months before lymphodepletion.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Participants must have adequate renal, cardiac, hepatic, pulmonary and bone marrow function as defined by the protocol.

Exclusion criteria:

1. Diagnosis of acute promyelocytic leukemia.
2. Has received or plans to receive any of the excluded therapy/treatment within the specified timeframe before lymphodepleting chemotherapy as defined by the protocol.
3. Prior allogeneic HSCT within 3 months of signing informed consent form (ICF) or with ongoing requirement for systemic graft-versus-host therapy.
4. Active central nervous system (CNS) involvement.
5. History of malignancy other than non-melanoma skin cancer or carcinoma in situ (eg. cervix, bladder, breast) low grade prostate cancer without treatment requirement unless in remission without treatment for ≥2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to 1 month
Maximum Tolerated Dose (MTD) of GDX012 | Up to 1 month
Number of Participants With Adverse Events (AEs) | Up to 14 months
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.

SECONDARY OUTCOMES:
Number of Participants With Disease Response | Up to 14 months
  Disease response includes participants achieving complete response [CR] complete response with incomplete hematologic recovery [CRi] (complete response with partial hematologic recovery [CRh] morphological leukemia-free state [MLFS] or partial response [PR] (based on 2022 European Leukemia Net [ELN] response criteria for AML after GDX012 administration.
Number of Participants With Measurable Residual Disease (MRD) Negative Status as Determined by Flow Cytometry | Up to 14 months
Duration of Response (DOR) | Up to 14 months
  DOR is defined as the time from the date of first documented CR, CRh, or CRi to the date of relapse or death.
Event-free Survival (EFS) | Up to 14 months
  EFS is defined as the time from the date of the first GDX012 administration to the date of treatment failure, relapse or death, whichever comes first.
Overall Survival (OS) | Up to 14 months
  OS is defined as the time from the date of the first GDX012 administration to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- United States (10):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Sarah Cannon/CBCI, Denver, Colorado
  - Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Thomas Jefferson University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Tri-Star BMT/Sarah Cannon Nashville, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- National Cancer Center Hospital East, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/fb2158ec7a43459e??page=1&idFilter=TAK-012-1501